CLINICAL TRIAL: NCT05488899
Title: Ultra Low Iodine Loaded Spectral CT Angiography (CTA) of the Aorta and Lower Limb: A Randomized Controlled Trial
Brief Title: Ultra Low Iodine Loaded Spectral CT Angiography (CTA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: Oslo Metropolitan University (Other)
Responsible Party: Principal Investigator, Peter Maehre Lauritzen, Researcher, Radiologist, PhD, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2018_070
Record Dates: First submitted 2022-06-21; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Peripheral Arterial Disease; Renal Insufficiency
Keywords: Computed Tomography Angiography; Contrast Media
MeSH Terms: conditions — Peripheral Arterial Disease; Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: RCT: Patients assigned to study or control group
Who Masked: Participant
Masking Description: Participants are not informed of which arm they are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Half iodine - Spectral CT group (Experimental): Patients receive half dosage of iodine contrast agent, and Spectral CT acquisition with Virtual Monoenergetic Images at 40 and 50 kiloelectronVolts (keV).
  Interventions: Diagnostic Test: Half iodine Spectral CT
- Standard iodine - Conventional CT (Active Comparator): Patients receive standard dosage of iodine contrast agent, and conventional 120 kiloVolts (kV) polychromatic CT images
  Interventions: Diagnostic Test: Standard iodine conventional CT

INTERVENTIONS:
Diagnostic Test: Half iodine Spectral CT — Patients receive half dosage of iodine contrast agent, and Spectral CT acquisition with Virtual Monoenergetic Images at 40 and 50 keV.
  Arms: Half iodine - Spectral CT group
Diagnostic Test: Standard iodine conventional CT — Patients receive standard dosage of iodine contrast agent, and conventional 120 kv Polychromatic CT acquisition.
  Arms: Standard iodine - Conventional CT

SUMMARY:
The objectives of this study are:

Evaluation of ultra-low iodine load CTA protocols of the aorta and lower extremities.

To investigate whether dual-layer in combination with with virtual monoenergetic imaging (VMI) allows for reduction of contrast medium (CM) in CTA of the aorta and lower limbs i with sustained objective and subjective image quality parameters.

DETAILED DESCRIPTION:
CT angiography (CTA) of the aorta and the lower limb is one of the most important tools for diagnostic, evaluation of the severity of the peripheral arterial disease, decision making, treatment planning and follow-up; but usually requires the use of iodine contrast medium.

Due to the high prevalence of renal impairment (eGFR < 90 ml/min/1.73m) in the elderly hospitalized population (more than 90% among inpatients aged over 60 years) contrast-medium-induced nephropathy is a major concern in this population.

The recently introduced spectral CT technique utilizes x-rays covering a spectrum of energy-levels as opposed to conventional CT in which x-rays are set to one specific energy level.

This technology offers many possibilities, such as "boosting" the x-ray contrast effect of iodine. This improves the vascular enhancement of the contrast medium using low-energy, virtual monoenergetic imaging (VNI).

The objectives of this study are:

Evaluation of ultra-low iodine load CTA protocols of the aorta and lower extremities.

To investigate whether dual-layer in combination with with virtual monoenergetic imaging (VMI) allows for reduction of contrast medium (CM) in CTA of the aorta and lower limbs i with sustained objective and subjective image quality parameters.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients and outpatients with kidney function (eGFR) allowing for safe administration of standard contrast dose (as calculated with the OmniVis calculator).
* Patients with clinical suspicion of disease of the aorta and/or arteries in the lower limb.
* Referral to CTA diagnosis, treatment planning or follow-up.

Exclusion Criteria:

* Iodine contrast medium allergy
* Age < 18 years
* Lack of informed consent
* Critical ischemia of the lower extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Mean arterial attenuation | Measured on CT images acquired at time of inclusion
  Attenuation (x-ray density) is measured in Hounsfield units (HU) digitally by placing a "region of interest" (ROI) circle in the Aorta, common iliac-, femoral- and popliteal arteries on the CT images acquired at the time of inclusion.

SECONDARY OUTCOMES:
Subjective examination quality | Rated on CT images acquired at time of inclusion
  Examination quality rated by interventional radiologists on a 4-point scale at the anatomic levels: aorta, common iliac, femoral, popliteal- and calf arteries.
  Subjective examination quality rating scale:
  1. (best) - Excellent: The demarcation of the vessel lumen is excellent, more than sufficient for confident diagnosis or exclusion of stenosis or occlusion.
  2. - Good: The demarcation of the vessel lumen is sufficient for confident diagnosis or exclusion of stenosis or occlusion.
  3. - Adequate: The demarcation of the vessel lumen is adequate for diagnosis or exclusion of stenosis or occlusion, but with limited confidence.
  4. (worst) - Non-diagnostic: There is insufficient demarcation of the vessel lumen for diagnosis or exclusion of stenosis or occlusion.
Rate of diagnostic quality angiography | Measured on images acquired at time of inclusion
  Based on measurements of attenuation in the aorta, common iliac-, femoral- and popliteal arteries. Diagnostic quality defined as arterial attenuation >200 Hounsfield units (HU)

OTHER OUTCOMES:
Image noise | Measured on CT-images acquired at time of inclusion
  Image noise was defined as the standard deviation of arterial attenuation measurements (see outcome 1) measured in HU digitally by placing a ROI on the CT-images in the aorta, common iliac-, femoral- and popliteal arteries.
Contrast to noise ratio (CNR) | Measured on CT-images acquired at time of inclusion
  Contrast to noise ratio was defined as: (Arterial attenuation - Background attenuation) / Image noise
  Arterial attenuation: (see outcome 1) measured in HU digitally by placing a ROI on the CT-images in the aorta, common iliac-, femoral- and popliteal arteries.
  Background attenuation: defined as attenuation in muscle measured in HU digitally by placing an identical size ROI on the CT-images in muscle tissue at the same anatomical levels as the arterial measurements.
  Image noise: see outcome 4
Signal to noise ratio (SNR) | Measured on CT-images acquired at time of inclusion
  Signal to noise ratio was defined as: Arterial attenuation / Image noise
  Arterial attenuation: (see outcome 1) measured in HU digitally by placing a ROI on the CT-images in the aorta, common iliac-, femoral- and popliteal arteries.
  Image noise: see outcome 4

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Lauritzen, MD PhD, Principal Investigator — University Hospital, Akershus & Oslo University Hospital
Locations (1):
- Akershus University Hospital, Lørenskog, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kristiansen CH, Thomas O, Tran TT, Roy S, Hykkerud DL, Sanderud A, Geitung JT, Lauritzen PM. Halved contrast medium dose in lower limb dual-energy computed tomography angiography-a randomized controlled trial. Eur Radiol. 2023 Sep;33(9):6033-6044. doi: 10.1007/s00330-023-09575-3. Epub 2023 Apr 18. PMID 37071166

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT05488899/Prot_SAP_000.pdf